CLINICAL TRIAL: NCT03673202
Title: A Clinical, Non-intervention Study of the Cxbladder Urine Test for the Detection of Recurrent Urinary Tract Urothelial Carcinoma
Brief Title: The Cxbladder Rule-out of Recurrent Urothelial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre (Other)
Collaborators: Pacific Edge Limited (Industry)
Responsible Party: Principal Investigator, Dr. Jonathan Izawa, Primary Investigator, London Health Sciences Centre
Other Study IDs: Waiting
Record Dates: First submitted 2018-09-06; First posted 2018-09-17 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients urine specimen are analysed for the test; kept in storage for 10 years for potential future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UC monitoring patients: Patients undergoing investigative cystoscopy for the detection of urothelial carcinoma as part of a standard-of-care schedule of investigations. All patients will have urine samples taken and analyzed for urine cytology and Cxbladder. No results for any tests under evaluation in this study are provided to the clinician for diagnostic purposes.
  Interventions: Diagnostic Test: Cx bladder Monitor test

INTERVENTIONS:
Diagnostic Test: Cx bladder Monitor test — Cxbladder Monitor is a non-invasive UC detection test measuring five messenger RNA (mRNA) biomarkers present at elevated levels in patients presenting with urothelial carcinoma and also two clinical variables (whether the previous tumor was primary or recurrent and the time since the previous tumor was resected).

SUMMARY:
This observational study is designed to collect urine and relevant clinical information from patients who have a known diagnosis of bladder cancer and currently on clinically driven surveillance. The study aims to compare the urine test to the flexible cystoscopy procedure (which the patient is already scheduled).

DETAILED DESCRIPTION:
There are approximately 360,000 new cases of bladder cancer diagnosed globally each year. In addition, this disease is responsible for 145,000 deaths annually (Parkin et al 2005). Treatments for this cancer range from transurethral resection of the bladder tumor (TURBT) for low stage, non-invasive tumors, to the more drastic option of radical cystectomy with pelvic lymph node dissection for those tumors that are found to have invaded into the muscularis propria (Parekh et al 2006). Currently, the standard of care for diagnosing bladder cancer involves a combination of flexible cystoscopy and urine cytology, which is usually performed after the patient presents with episodes of gross hematuria. Following these evaluations, if evidence exists that warrants further investigation for bladder cancer a TURBT is performed and accurate staging and grading of the tumor can occur (O'Sullivan et al 2012). For those patients who have localized disease and have bladder preservation therapies, long term surveillance (in high grade disease this is life-long) is required to monitor for recurrence of tumor (Sylvester et al 2006). While cystoscopy has proven to be an accurate tool (sensitivity 80%) in the surveillance of bladder cancer, it is nonetheless a highly invasive procedure (Jocham et al 2008). In addition, urine cytology, which has served as the traditional adjunct to cystoscopy operates with a modest degree of sensitivity and therefore potential to deliver false negatives where malignant cells are not seen and false positives for bladder cancer in patients with an acute or chronically inflamed urothlelium (Grossman et al 2005). This leaves room for the development of a diagnostic test that is able to deliver results with the specificity of cystoscopy but without the potential for false negatives seen with urine cytology.

Recently, studies have shown that certain genetic markers exist that accompany the occurrence of bladder cancer and can accurately discriminate between bladder tumors and normal tissue. These genetic markers also show promise in being able to deliver additional information regarding the disease state of this cancer, such the stage and grade of the tumor (Dyrskjot et al 2003; Dyrskjot et al 2005; Thykjaer et al 2001). The informative nature of these mRNA expression profiles, along with the frequency with which tumor exfoliation into the urine occurs, has led to the development of a urine-based test that has the potential to diagnose and stratify bladder cancer. This urine test, known as Cxbladder Monitor, was developed by Pacific Edge Limited and is able to perform a combinatory analysis of the expression profiles of five genetic biomarkers (IGF, HOXA, MDK, CDC and IL8R gene expression) and two clinical variables (whether the previous tumor was primary or recurrent and the time since the previous tumor was resected). This test has the potential, with further testing, to produce a consolidated diagnostic score that is able to accurately risk stratify a given patient for recurrence of bladder cancer based on tumor characteristics. The five genetic markers include CDC2 (a gene involved in cell cycle activity and DNA synthesis) (O'Sullivan et al 2012), HOXA13 (transcription factor involved in morphogenesis and differentiation of the genitourinary tract) (Scott et al 2005), IGFBP5 (affects processes such as such as development, differentiation, and cellular survival) (Beattie et al 2006), MDK (a heparin binding growth factor expressed during embryogenesis) (Kadomatsu et al 2004), and CXCR2 which is expressed in neutrophils and is increased in non-malignant, inflammatory conditions. This marker is essential as it is helpful in reducing the risk of false positive results in patients with an inflamed urothelium (O'Sullivan et al 2012). The Cxbladder test is able to take into account the expression of all these relevant genetic markers and analyze their expression profiles and interactions via a 2 way linear discriminate algorithm to form a score that is able to predict the recurrence of bladder cancer. The success of these preliminary studies with Cxbladder show that it has a strong potential to be used as a alternate to urine cytology and challenge cytology's routine accompaniment to cystoscopy. More importantly, the use of Cxbladder in the surveillance patient has the potential to decrease the frequency with which cystoscopy would need to be performed, adjudicate equivocal cystoscopy and cytology atypia.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is undergoing investigative cystoscopies for the monitoring of recurrence of urinary tract UC at intervals prescribed by the clinical practitioner
2. Patients on an "all-comers" basis
3. Positive diagnosis for primary or recurrent bladder tumour within the past 5 years
4. Able provide a voided urine sample of the required minimum volume
5. Able to give written consent
6. Able and willing to comply with study requirements
7. Aged 18 years or older

Exclusion Criteria:

1. Prior genitourinary manipulation (flexible or rigid cystoscopy / catheterisation, urethral dilation) in the 14 days before urine collection,
2. Patients who had exposure to intravesical BCG, had completed induction BCG but without a subsequent clear cystoscopy
3. Recent history of glomerulonephritis, nephrosis or other renal inflammatory disorders,
4. Recent history of pyelonephritis
5. Total cystectomy of the bladder, neo bladders and illeal conduits
6. Previous muscle invasive bladder tumour (pT2 or greater)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing flexible cystoscopy on a clinically determined surveillance schedule who have been previous diagnosed with bladder cancer are eligible. These patients are recruited prior to their investigation, and a urine sample collected. The patients clinical events are then followed (observed) for 12 months following the urine sample collection.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with bladder cancer who are correctly identified as having cancer (true positives) and no cancer (true negatives) by the Cxbladder test. | 24 months
  To validate the Performance Characteristics (sensitivity, area under the ROC curve, positive and negative predictive values and test negative rate) of the Cxbladder for the detection of recurrent UC in the absence of inflammation in patients with a recent history of urinary tract UC who have been treated according to standard practice and are undergoing routine investigative cystoscopy. The gold standard for determination of clinical truth is cystoscopy confirmed by pathology, plus any follow up investigations relating to the current visit.

SECONDARY OUTCOMES:
Detection rates of Cx bladder test | 24 months
  To define and the validate the Performance Characteristics of the Cxbladder for the detection of recurrent UC in local population patients with a recent history of urinary tract UC who have been treated according to standard practice and are undergoing routine investigative cystoscopy
Comparison of Cxbladder theoretical capacity to reduce use of flexible cystoscopy for the monitoring for recurrence of urothelial carcinoma | 24 months
  To estimate the theoretical clinical outcome of patients under the Standard Of Care tested with Cxbladder before investigative cystoscopy to determine the true proportion requiring cystoscopy and follow up and thereby determining the potential of Cxbladder for reducing the cystoscopy burden on patients undergoing monitoring for recurrence
Comparison of the Cxbladder test and cytology test performance on the same sample | 12 months
  Performance characteristics (sensitivity, specificity, rule-out rate, PPV and NPV) of the Cxbladder and urine cytology on the same voided urine sample.
Performance of Cxbladder test in atypical findings of cytology and cystoscopy | 24 months
  To compare and contrast atypical cytology and / or equivocal cystoscopy with the performance characteristics of Cxbladder signatures
Examine urinary microbiome profile in patients with urothelial cancer | 24 months
  Compare differences in microbiome profiles in patients with urothelial cancer and those without

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Izawa, MD, Principal Investigator — Schulich School of Medicine and Dentistry
Locations (1):
- Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Parekh DJ, Bochner BH, Dalbagni G. Superficial and muscle-invasive bladder cancer: principles of management for outcomes assessments. J Clin Oncol. 2006 Dec 10;24(35):5519-27. doi: 10.1200/JCO.2006.08.5431. PMID 17158537
- [Background] O'Sullivan P, Sharples K, Dalphin M, Davidson P, Gilling P, Cambridge L, Harvey J, Toro T, Giles N, Luxmanan C, Alves CF, Yoon HS, Hinder V, Masters J, Kennedy-Smith A, Beaven T, Guilford PJ. A multigene urine test for the detection and stratification of bladder cancer in patients presenting with hematuria. J Urol. 2012 Sep;188(3):741-7. doi: 10.1016/j.juro.2012.05.003. Epub 2012 Jul 19. PMID 22818138
- [Background] Sylvester RJ, van der Meijden AP, Oosterlinck W, Witjes JA, Bouffioux C, Denis L, Newling DW, Kurth K. Predicting recurrence and progression in individual patients with stage Ta T1 bladder cancer using EORTC risk tables: a combined analysis of 2596 patients from seven EORTC trials. Eur Urol. 2006 Mar;49(3):466-5; discussion 475-7. doi: 10.1016/j.eururo.2005.12.031. Epub 2006 Jan 17. PMID 16442208
- [Background] Jocham D, Stepp H, Waidelich R. Photodynamic diagnosis in urology: state-of-the-art. Eur Urol. 2008 Jun;53(6):1138-48. doi: 10.1016/j.eururo.2007.11.048. Epub 2007 Dec 10. PMID 18096307
- [Background] Grossman HB, Messing E, Soloway M, Tomera K, Katz G, Berger Y, Shen Y. Detection of bladder cancer using a point-of-care proteomic assay. JAMA. 2005 Feb 16;293(7):810-6. doi: 10.1001/jama.293.7.810. PMID 15713770
- [Background] Dyrskjot L, Thykjaer T, Kruhoffer M, Jensen JL, Marcussen N, Hamilton-Dutoit S, Wolf H, Orntoft TF. Identifying distinct classes of bladder carcinoma using microarrays. Nat Genet. 2003 Jan;33(1):90-6. doi: 10.1038/ng1061. Epub 2002 Dec 9. PMID 12469123
- [Background] Dyrskjot L, Zieger K, Kruhoffer M, Thykjaer T, Jensen JL, Primdahl H, Aziz N, Marcussen N, Moller K, Orntoft TF. A molecular signature in superficial bladder carcinoma predicts clinical outcome. Clin Cancer Res. 2005 Jun 1;11(11):4029-36. doi: 10.1158/1078-0432.CCR-04-2095. PMID 15930337
- [Background] Thykjaer T, Workman C, Kruhoffer M, Demtroder K, Wolf H, Andersen LD, Frederiksen CM, Knudsen S, Orntoft TF. Identification of gene expression patterns in superficial and invasive human bladder cancer. Cancer Res. 2001 Mar 15;61(6):2492-9. PMID 11289120
- [Background] Scott V, Morgan EA, Stadler HS. Genitourinary functions of Hoxa13 and Hoxd13. J Biochem. 2005 Jun;137(6):671-6. doi: 10.1093/jb/mvi086. PMID 16002988
- [Background] Beattie J, Allan GJ, Lochrie JD, Flint DJ. Insulin-like growth factor-binding protein-5 (IGFBP-5): a critical member of the IGF axis. Biochem J. 2006 Apr 1;395(1):1-19. doi: 10.1042/BJ20060086. PMID 16526944
- [Background] Kadomatsu K, Muramatsu T. Midkine and pleiotrophin in neural development and cancer. Cancer Lett. 2004 Feb 20;204(2):127-43. doi: 10.1016/S0304-3835(03)00450-6. PMID 15013213